CLINICAL TRIAL: NCT05800821
Title: Prediction of Cerebral Hyperperfusion Syndrome After Carotid Revascularization Using Deep Learning
Status: Recruiting | Type: Observational
Sponsor: State Institution "Republican Scientific and Practical Center" Cardiology, Belarus (Other)
Responsible Party: Principal Investigator, Dr. Ivan Maiseyenka, Principal Investigator, Vascular Surgery Research Laboratory, State Institution "Republican Scientific and Practical Center" Cardiology, Belarus
Other Study IDs: 455; 20251402/497 (Other: State Committee on Science and Technology)
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Carotid Artery Diseases; Carotid Atherosclerosis; Carotid Artery Stenosis; Cerebral Hyperperfusion Syndrome
Keywords: Cerebral Hyperperfusion Syndrome; Carotid Stenosis; Stroke; Deep Learning
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Reduced Cerebrovascular Reserve
  Interventions: Procedure: Carotid revascularization
- Patients with Sufficient Cerebrovascular Reserve
  Interventions: Procedure: Carotid revascularization

INTERVENTIONS:
Procedure: Carotid revascularization — Carotid revascularization

SUMMARY:
Cerebral hyperperfusion syndrome (CHS) was initially described as a clinical complication following carotid endarterectomy (CEA), but it may occur after both CEA and carotid artery stenting. It is characterised by throbbing ipsilateral frontotemporal or periorbital headache, and sometimes diffuse headache, eye and facial pain, vomiting, confusion, macular oedema, visual disturbances, focal motor seizures with frequent secondary generalisation, focal neurological deficits, and intracerebral or subarachnoid haemorrhage.

Knowledge of CHS among physicians remains limited. Most studies report an incidence of 1-3% after carotid endarterectomy. CHS is most common in patients with increases of more than 100% in cerebral perfusion compared with baseline after carotid revascularization, and is rare in patients with perfusion increases of less than 100% compared with baseline.

The pathophysiological mechanism of CHS is only partially understood. The chronic low-flow state induced by severe carotid disease results in compensatory dilation of cerebral vessels distal to the stenosis, as part of the normal autoregulatory response to maintain adequate cerebral blood flow (CBF). In this chronically dilated state, the vessels lose their ability to autoregulate vascular resistance in response to changes in blood pressure. Dysautoregulation has been shown to be proportional to the duration and severity of chronic hypoperfusion. After revascularization and reperfusion, impaired cerebral autoregulation may contribute to a cascade of intracranial microcirculatory changes, with an inability to respond adequately to the augmentation of CBF following carotid recanalization.

Although most patients present with mild symptoms and signs, progression to severe and life-threatening complications can occur if CHS is not recognised and treated promptly. Because CHS is diagnosed on the basis of several non-specific signs and symptoms, patients may be misdiagnosed as having one of the better-known causes of perioperative complications, such as thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 80 years.
2. Occlusive-stenotic lesion of the carotid arteries with indications for carotid revascularization.

Exclusion Criteria:

1. Systemic vasculitis.
2. Cerebral vessel aneurysms.
3. Arteriovenous malformation of the brain.
4. Primary brain tumor (including metastatic lesions).
5. Epilepsy.
6. History of traumatic brain injury.
7. Demyelinating diseases of the central nervous system.
8. History of neuroinfection.
9. Atrial fibrillation.
10. Frequent supraventricular or ventricular extrasystoles.
11. Chronic heart failure with left ventricular ejection fraction less than 40%.
12. Chronic kidney disease with estimated glomerular filtration rate less than 45 mL/min/1.73 m².
13. Presence of an implanted cardioverter-defibrillator or pacemaker.
14. Presence of contraindications to the medical use of iodine-containing radiographic contrast agents.
15. Patient's unwillingness to continue participating in the study.
16. Absence of a temporal acoustic window for transcranial Doppler ultrasonography.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo carotid revascularization procedures
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2028-05-03 (Estimated); Study Completion 2030-05-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Cerebral Hyperperfusion Syndrome | Occurrence of symptoms within 30 postoperative days
  The diagnosis of cerebral hyperperfusion syndrome will be based on the following criteria:
  1. Appearance of symptoms within 1 month after surgery.
  2. First-time unilateral headache, convulsions, hemiparesis/hemiplegia, visual disturbances, ataxia, Glasgow Coma Scale score < 15 points, aphasia, or signs of cerebral edema or intracerebral hemorrhage.
  3. Symptoms of "luxury perfusion syndrome" occurring within the first 24-48 hours after restoration of blood flow through the internal carotid artery.
  4. Increase in cerebral blood flow in the middle cerebral artery > 100% compared with the preoperative value, measured by transcranial Doppler ultrasonography.
  5. Exclusion of differential diagnoses, including hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome, and reversible cerebral vasoconstriction syndrome.
  6. Neurological symptoms occurring in the context of high blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- State Institution "Republican Scientific and Practical Center "Cardiology", Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided